CLINICAL TRIAL: NCT06902441
Title: Impact of Androgen Receptor Signaling Inhibitors on Cardiovascular Events in Prostate Cancer: a Pharmacoepidemiology Study Using the French Health Care Claims Database
Brief Title: Impact of New Hormonotherapy Drugs in Prostatic Cancer on the Risk of Cardiovascular Events : a Pharmacoepidemiology Study Using the French Health Care Claims Database
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 20250318
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Androgen Receptor Signaling Inhibitors; Cardiovascular toxicity; Hormonotherapy; Pharmacoepidemiology
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Apalutamide: Data collected about patients treated with Apalutamide
- Abiraterone Acetate: Data collected about patients treated with Abiraterone Acetate
- Enzalutamide: Data collected about patients treated with Enzalutamide

SUMMARY:
In prostate cancer, whether advanced or localized, hormone therapy is a key treatment. These therapies work by lowering male hormone levels to slow the growth of cancer.

More recently, a new group of medications called Androgen Receptor Signaling Inhibitors (ARSIs) has been introduced. These drugs are used alongside standard hormone therapy and are now prescribed for both advanced and high-risk localized prostate cancer.

There are two main types of ARSIs: abiraterone acetate, which blocks the body from making androgens, and enzalutamide, apalutamide, and darolutamide, which stop cancer cells from using these hormones. Doctors choose among them based on individual patient needs, as no one drug has been clearly shown to be better than the others. These treatments have significantly improved survival for many patients.

However, research shows that 30% of men with prostate cancer die from heart-related issues-a higher rate than in the general population. It's important to better understand how these treatments might be linked to heart risks.

One study found that all ARSIs increase the risk of serious heart problems. However, it did not take into account whether patients already had heart conditions, even though previous heart issues are known to increase the risk with certain drugs like abiraterone and enzalutamide.

That's why we're conducting a study using a large real-world database to compare the heart risks of abiraterone, enzalutamide, and apalutamide. We will take into account both patients' existing heart conditions and how long they were on treatment.

DETAILED DESCRIPTION:
In prostate cancer, both in metastatic settings and in many localized cases, androgen suppression via Gonadotropin-Releasing Hormone (GnRH) agonists or antagonists remains the cornerstone of treatment. These androgen deprivation therapies (ADT) aim to reduce circulating androgen levels.

In recent years, Androgen Receptor Signaling Inhibitors (ARSIs) have emerged and are now prescribed in combination with ADT. These treatments have broad indications in metastatic settings and are also increasingly used in localized high-risk prostate cancer.

A conventional distinction is made between abiraterone acetate-a selective inhibitor of androgen synthesis that blocks CYP17-and other ARSIs that inhibit the androgen receptor, namely enzalutamide, apalutamide, and darolutamide. The indications for these treatments are often similar, with no clear evidence supporting the superiority of one over another. For instance, in synchronous metastatic hormone-sensitive prostate cancer, when treated with ARSIs combined with ADT, clinicians may choose between abiraterone acetate, apalutamide, or enzalutamide. Thus, the safety profile of these agents plays a crucial role in therapeutic decision-making. These next-generation hormonal therapies have significantly improved patient survival.

However, when examining causes of death among patients with prostate cancer, studies have shown that 30% of deaths are due to cardiovascular causes, with an excess risk compared to the general population. It is therefore essential to investigate these cardiovascular events and their associations with the treatments administered.

One meta-analysis identified an increased risk of high-grade cardiovascular toxicities associated with all next-generation hormonal therapies (HR 1.75; 95% CI: 1.50-2.04). This excess risk was observed for each ARSI individually. However, the meta-analysis could not account for patients' cardiovascular history, despite demonstrated associations between pre-existing cardiovascular conditions and the risk of cardiovascular toxicity with abiraterone acetate and enzalutamide.

For these reasons, we aimed to compare cardiovascular toxicities associated with abiraterone, enzalutamide, and apalutamide using a large real-world database, taking into account pre-existing cardiovascular comorbidities as well as treatment exposure duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients had to begin a treatment with Enzalutamide, Abiraterone or Apalutamide between the 01-01-2018 and the 31-12-2022
* Patients must have a unique ID in the database, to be able to link the data

Exclusion Criteria:

* Previous treatment with another novel androgen receptor signaling inhibitors
* Patients were excluded if they began a chemotherapy treatment in the 6 weeks following the beginning of Androgen Receptor Signaling Inhibitors (ARSI)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostatic cancer treated with an ARSI amoung Abiraterone Acetate, Enzalutamide or Apalutamide.
Sampling Method: Non-Probability Sample
Enrollment: 52000 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Risk of hospitalization for cardiovascular cause | From the beginning of the ARSI to the first date among : death, end of hormonotherapy, study endpoint date (31-12-2023) or outcome
  The primary objective of this study was to compare the risk of hospitalization for cardiovascular reasons among the different Androgen Receptor Signaling Inhibitors (ARSI). This outcome was evaluated by the occurrence of a hospitalization for one of these reasons as the principal diagnosis.

SECONDARY OUTCOMES:
Risk of hospitalization for hearth failure | From the beginning of the ARSI to the first date among : death, end of hormonotherapy, study endpoint date (31-12-2023) or outcome
  One of the secondary objective of this study was to compare the risk of hospitalization for heart failure amoung the different Androgen Receptor Signaling Inhibitors (ARSI). This outcome was evaluated by the occurrence of a hospitalization for heart failure as the principal diagnosis (International Classification of Diseases, 10th Edition; code I50).
Risk of hospitalization for atrial fibrillation | From the beginning of the ARSI to the first date among : death, end of hormonotherapy, study endpoint date (31-12-2023) or outcome
  One of the secondary objective of this study was to compare the risk of hospitalization for atrial fibrillation or flutter amoung the different Androgen Receptor Signaling Inhibitors (ARSI). This outcome was evaluated by the occurrence of a hospitalization for atrial fibrillation or flutter as the principal diagnosis (International Classification of Diseases, 10th Edition; code I48).
Risk of hospitalization for ischemic heart disease | From the beginning of the ARSI to the first date among : death, end of hormonotherapy, study endpoint date (31-12-2023) or outcome
  One of the secondary objective of this study was to compare the risk of hospitalization for ischemic heart disease amoung the different Androgen Receptor Signaling Inhibitors (ARSI). This outcome was evaluated by the occurrence of a hospitalization for ischemic heart disease as the principal diagnosis (International Classification of Diseases, 10th Edition; code I20-I25).
Risk of hospitalization for hypertensive disease | From the beginning of the ARSI to the first date among : death, end of hormonotherapy, study endpoint date (31-12-2023) or outcome
  One of the secondary objective of this study was to compare the risk of hospitalization for hypertensive disease amoung the different Androgen Receptor Signaling Inhibitors (ARSI). This outcome was evaluated by the occurrence of a hospitalization for hypertensive disease as the principal diagnosis (International Classification of Diseases, 10th Edition; code I10-I13; I15).
Risk of hospitalization for successfully resuscitated cardiac arrest | From the beginning of the ARSI to the first date among : death, end of hormonotherapy, study endpoint date (31-12-2023) or outcome
  One of the secondary objective of this study was to compare the risk of hospitalization for resuscitated cardiac arrest amoung the different Androgen Receptor Signaling Inhibitors (ARSI). This outcome was evaluated by the occurrence of a hospitalization for resuscitated cardiac arrest as the principal diagnosis (International Classification of Diseases, 10th Edition; code I50)
Risk of death | From the beginning of the ARSI to the first date among : death, end of hormonotherapy, study endpoint date (31-12-2023)
  Another secondary objective was to evaluate the risk of death under Androgen Receptor Signaling Inhibitors (ARSI) treatment. This objective was assessed by the occurrence of death, regardless of the cause.
Risk of new registration for long term illness | From the beginning of the ARSI to the first date among : death, end of hormonotherapy, study endpoint date (31-12-2023) or outcome
  Finally, a further secondary objective was to compare the risk of a new registration for long-term illness due to cardiovascular reasons, according to the Androgen Receptor Signaling Inhibitors (ARSI) used.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baser O, Samayoa G, Dwivedi A, AlSaleh S, Cigdem B, Kizilkaya E. Cardiovascular events among patients with prostate cancer treated with abiraterone and enzalutamide. Acta Oncol. 2024 Apr 9;63:137-146. doi: 10.2340/1651-226X.2024.20337. PMID 38591349
- [Background] Lu-Yao G, Nikita N, Keith SW, Nightingale G, Gandhi K, Hegarty SE, Rebbeck TR, Chapman A, Kantoff PW, Cullen J, Gomella L, Kelly WK. Mortality and Hospitalization Risk Following Oral Androgen Signaling Inhibitors Among Men with Advanced Prostate Cancer by Pre-existing Cardiovascular Comorbidities. Eur Urol. 2020 Feb;77(2):158-166. doi: 10.1016/j.eururo.2019.07.031. Epub 2019 Aug 13. PMID 31420248
- [Background] El-Taji O, Taktak S, Jones C, Brown M, Clarke N, Sachdeva A. Cardiovascular Events and Androgen Receptor Signaling Inhibitors in Advanced Prostate Cancer: A Systematic Review and Meta-Analysis. JAMA Oncol. 2024 Jul 1;10(7):874-884. doi: 10.1001/jamaoncol.2024.1549. PMID 38842801
- [Background] Ye Y, Zheng Y, Miao Q, Ruan H, Zhang X. Causes of Death Among Prostate Cancer Patients Aged 40 Years and Older in the United States. Front Oncol. 2022 Jul 1;12:914875. doi: 10.3389/fonc.2022.914875. eCollection 2022. PMID 35847902
- [Background] Ploussard G, Baboudjian M, Barret E, Brureau L, Fiard G, Fromont G, Olivier J, Dariane C, Mathieu R, Rozet F, Peyrottes A, Roubaud G, Renard-Penna R, Sargos P, Supiot S, Turpin L, Roupret M; Comite de Cancerologie de l'Association Francaise d'Urologie, Groupe Prostate, Maison de l'Urologie. French AFU Cancer Committee Guidelines - Update 2024-2026: Prostate cancer - Diagnosis and management of localised disease. Fr J Urol. 2024 Nov;34(12):102717. doi: 10.1016/j.fjurol.2024.102717. PMID 39581668